CLINICAL TRIAL: NCT01451476
Title: Human Skin Aging: Clinical Parameters and Gene Expression Profiling
Acronym: GEP
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anne Chang, instructor, Stanford University
Other Study IDs: HSA_GEP; 003 (Other Grant/Funding Number: NuSkin International)
Record Dates: First submitted 2011-10-11; First posted 2011-10-13 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Ageing
Keywords: Ageing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and skin samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy females aged >=18: Healthy female volunteers of skin type I or II

SUMMARY:
Skin aging is a complex process involving genetic and environmental factors. The investigators hope to learn more about how human genes and their function can contribute to skin aging and human health.

DETAILED DESCRIPTION:
This study includes answering a survey on prior sun exposures, donating two small pieces of skin (4mm each), one blood draw, complexion analysis, photographs, and non-invasive tests such as skin surface lipid analysis. Your blood and tissue will be sent for DNA analysis and gene expression profiling.

ELIGIBILITY:
Inclusion Criteria:

* healthy female, age 18 or older,
* Fitzpatrick type 1 or 2 skin,
* able to read and understand written consent form,
* body mass index normal or overweight range,
* willing to take blood tests and donate skin samples

Exclusion Criteria:

* pregnant or lactating,
* history of cosmetic surgery affecting the face,
* use of prescription anti-aging medications for 2 weeks prior to study,
* use of dietary supplements for 2 weeks prior to study, use of tanning beds or excessive light exposure (>2 hours) in the past 2 weeks,
* medical conditions which at the discretion of the investigator will have significant impact on ability to judge subjects' skin characteristics and age, sunless tanner use in past 2 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy females age 18 or older
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2010-05; Primary Completion 2015-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Assessment of age related gene expression changes in skin | Cross sectional

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Lane, MD, Principal Investigator — Stanford University; Anne Chang, MD, Study Director — Stanford University
Locations (1):
- Stanford Dermatology, Redwood City, California, United States

REFERENCES:
- [Result] Xu J, Spitale RC, Guan L, Flynn RA, Torre EA, Li R, Raber I, Qu K, Kern D, Knaggs HE, Chang HY, Chang AL. Novel Gene Expression Profile of Women with Intrinsic Skin Youthfulness by Whole Transcriptome Sequencing. PLoS One. 2016 Nov 9;11(11):e0165913. doi: 10.1371/journal.pone.0165913. eCollection 2016. PMID 27829007